CLINICAL TRIAL: NCT02764814
Title: In Vivo Confocal Microscopic Analysis of Corneal Nerve Changes After ProKera Slim® for Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: P014-03
Record Dates: First submitted 2016-04-25; First posted 2016-05-06 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): subjects receiving cryopreserved amniotic membrane
  Interventions: Other: Cryopreserved amniotic membrane
- Control (No Intervention): no intervention

INTERVENTIONS:
Other: Cryopreserved amniotic membrane — subjects will receive cryopreserved amniotic membrane
  Other Names: ProKera Slim
  Arms: Treatment

SUMMARY:
Prospective controlled pilot study to compare the outcome of ProKera® (PK) and conventional treatment in patients with moderate to severe Dry Eye Disease (DED)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe DED (Grade 2-4 DEWS)
* Age range: 21 years and older.
* Both genders and all ethnic groups comparable with the local community.
* Subjects able to understand and willing to sign a written informed consent.
* Subjects able and willing to cooperate with investigational plan.
* Subjects able and willing to complete postoperative follow-up.

Exclusion Criteria:

* Symblepharon or lid abnormality preventing ProKera placement.
* Ocular infection within 14 days prior to study entry.
* Active ocular allergies.
* Previous ocular surgery or injury within 3 months before enrollment.
* Previous brain surgery, or Trigeminal nerve damage.
* Other conditions that may affect corneal nerves such as diabetes, thyroid disorders.
* Contact lens wearers.
* Pregnancy or subject expecting to be pregnant.
* Inability or unwillingness of subject to give written informed consent.
* Subjects with known intolerance to PK.
* Subjects use concomitant therapy that affects tear functions or ocular surface integrity.
* Subjects currently engaged in another clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Short-term efficacy in terms of corneal nerve regeneration | Change from Baseline to 1 month
  Assessed by corneal topography
Short-term efficacy in terms of ocular surface integrity | Change from Baseline to 1 month
  Assessed by in vivo confocal microscopy
Short-term efficacy in terms of corneal sensitivity | Change from Baseline to 1 month
Short-term efficacy in terms of ocular clinical symptoms | Change from Baseline to 1 month
  Assessed by SPEED questionnaire, pain score, and dry eye workshop grading

SECONDARY OUTCOMES:
Long-term efficacy in terms of corneal nerve regeneration | Change from Baseline to 3 month
  Assessed by corneal topography
Long-term efficacy in terms of ocular surface integrity | Change from Baseline to 3 month
  Assessed by in vivo confocal microscopy
Long-term efficacy in terms of corneal sensitivity | Change from Baseline to 3 month
Long-term efficacy in terms of ocular clinical symptoms | Change from Baseline to 3 month
  Assessed by SPEED questionnaire, pain score, and dry eye workshop grading

CONTACTS AND LOCATIONS:
Overall Officials: Thomas John, MD, Principal Investigator — Thomas John Vision Institute
Locations (1):
- Thomas John Vision Institute, P.C., Tinley Park, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] John T, Tighe S, Sheha H, Hamrah P, Salem ZM, Cheng AMS, Wang MX, Rock ND. Corneal Nerve Regeneration after Self-Retained Cryopreserved Amniotic Membrane in Dry Eye Disease. J Ophthalmol. 2017;2017:6404918. doi: 10.1155/2017/6404918. Epub 2017 Aug 15. PMID 28894606